CLINICAL TRIAL: NCT01644604
Title: The Clinical Study of Renal Denervation by MDT-2211 System in Patients With Uncontrolled Hypertension
Brief Title: Renal Denervation by MDT-2211 System in Patients With Uncontrolled Hypertension
Acronym: HTN-J
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT2-11-07
Record Dates: First submitted 2012-06-29; First posted 2012-07-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Uncontrolled Hypertension
Keywords: Hypertension; Vascular Diseases; Cardiovascular Diseases; Renal denervation
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal denervation (Experimental): Subjects are treated with the renal denervation procedure after randomization and are maintained on baseline anti-hypertensive medications.
  Interventions: Device: MDT-2211 Renal Denervation System
- Control Group (No Intervention): Subjects are maintained on baseline anti-hypertensive medications

INTERVENTIONS:
Device: MDT-2211 Renal Denervation System — A percutaneous system that delivers radiofrequency (RF) energy through the luminal surface of the renal artery.
  Arms: Renal denervation

SUMMARY:
The objective of this study is to demonstrate that the MDT-2211 renal denervation system is a safe and effective treatment for uncontrolled hypertension subjects despite treatment with 3 or more anti-hypertensive medications of different classes, of which one must be a diuretic, as best available antihypertensive therapy

DETAILED DESCRIPTION:
The HTN-J study is a multi-center, prospective, unblinded, randomized, controlled study of the safety and effectiveness of renal denervation in subjects with uncontrolled hypertension. Bilateral renal denervation will be performed using the MDT-2211 renal denervation system - a percutaneous system that delivers radiofrequency (RF) energy through the luminal surface of the renal artery.

ELIGIBILITY:
Inclusion Criteria:

* Individual is ≥ 20 and ≤ 80 years old at time of randomization.
* Individual is receiving a stable medication regimen including full tolerated doses of 3 or more anti-hypertensive medications of different classes, of which one must be a diuretic (with no changes for a minimum of 6 weeks prior to screening) that is expected to be maintained without changes for at least 6 months.
* Individual has an office systolic blood pressure (SBP) of ≥ 160 mmHg based on an average of 3 blood pressure readings measured at both an initial screening visit and a confirmatory screening visit
* Individual agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria highlights:

* Individual has an estimated glomerular filtration rate (eGFR) of < 45 mL/min/1.73 m2
* Individual has an Ambulatory Blood Pressure Monitoring (ABPM) 24 hour average SBP < 135 mmHg
* Individual has type 1 diabetes mellitus
* Individual requires chronic oxygen support or mechanical ventilation (e.g., tracheostomy, CPAP, BiPAP) other than nocturnal respiratory support for sleep apnea.
* Individual has primary pulmonary hypertension.
* Individual is pregnant, nursing or planning to be pregnant.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Office Systolic Blood Pressure | Baseline to 6 months post-randomization

SECONDARY OUTCOMES:
Incidence of Major Adverse Events (MAE) | Baseline through 1 month post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Kazuyuki Shimada, MD, Principal Investigator — New Oyama Municipal Hospital
Locations (17):
- Japan (17):
  - Hirosaki University School of Medicine & Hospital, Hirosaki-shi, Aomori
  - Chiba University Hospital, Chiba, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Higashi Takarazuka Satoh Hospital, Takarazuka, Hyōgo
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Yokohama Tobu Hospital, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Sakyo-ku, Kyoto
  - Osaka University Hospital, Suita-shi, Osaka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Mitsui Memorial Hospital, Chiyoda-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo

REFERENCES:
- [Derived] Kario K, Bhatt DL, Brar S, Cohen SA, Fahy M, Bakris GL. Effect of Catheter-Based Renal Denervation on Morning and Nocturnal Blood Pressure: Insights From SYMPLICITY HTN-3 and SYMPLICITY HTN-Japan. Hypertension. 2015 Dec;66(6):1130-7. doi: 10.1161/HYPERTENSIONAHA.115.06260. Epub 2015 Oct 5. PMID 26558819
- [Derived] Kario K, Ogawa H, Okumura K, Okura T, Saito S, Ueno T, Haskin R, Negoita M, Shimada K; SYMPLICITY HTN-Japan Investigators. SYMPLICITY HTN-Japan - First Randomized Controlled Trial of Catheter-Based Renal Denervation in Asian Patients -. Circ J. 2015;79(6):1222-9. doi: 10.1253/circj.CJ-15-0150. Epub 2015 Apr 24. PMID 25912693